CLINICAL TRIAL: NCT01974063
Title: Alternate Nicotine Delivery Systems and Airway Epithelial Biology
Status: Terminated | Type: Observational
Why Stopped: Grant Ended
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 1208012965; R01HL107882-02S1 (NIH)
Record Dates: First submitted 2012-12-20; First posted 2013-11-01 (Estimated); Last update posted 2018-05-03 (Actual); Status verified 2018-04

CONDITIONS: Smoking; Smoking Cessation
Keywords: Smoking; Smoking Cessation; Healthy Smoker; Shisha Smoker; Non-smoker
MeSH Terms: conditions — Smoking; Smoking Cessation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Analysis performed will be completed per the "Airway" (IRB#1204012331) protocol.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (5):
- A. Nonsmokers: Subjects have smoked <100 cigarettes or <10 shisha pipes per lifetime and whose urine nicotine <2 ng/mL and/or urine cotinine <5 ng/mL, at entry into the study.
- B.Current cigarette smokers: Defined by self-report and urine nicotine >30 ng/mL and/or urine cotinine >50 ng/ml.
- C. Current shisha smokers: Defined by self-report of smoking >4 pipes/wk and carboxyhemoglobin >2.5.
- D. smokers willing to quit: Defined by self-report and urine nicotine >30 ng/ml and/or urine cotinine >50 ng/ml. Subjects must be a current smoker willing to stop smoking. Subjects will stop smoking after the baseline bronchoscopy, and switch to taking a smoking cessation medication called varenicline. We will provide subjects with the smoking cessation medication as part of this study. They will also receive phone calls to help with smoking cessation counseling.
- E. Smokers switching to E-cigarettes: Defined by self-report and urine nicotine >30 ng/ml and/or urine cotinine >50 ng/ml. Must be willing to switch from tobacco cigarettes to electronic cigarettes. The switch will occur after the baseline bronchoscopy. The nicotine dose that will be given to each subject will be determined by the study physician based on the urine smoking metabolite test. It will be adjusted depending on whether the subject is a light smoker or heavy smoker (Light smoker defined as having either a urine nicotine value from 2ng/ml-1000ng/ml or a urine cotinine value from 5ng/ml-1000ng/ml. Heavy smoker is defined as having either a urine nicotine or cotinine value of over 1000ng/ml.) We will provide the subjects with the electronic cigarettes to use as part of this study.

SUMMARY:
Cigarette smoking evokes major changes in the biology of the airway epithelium, the cell population that takes the brunt of the stress of cigarette smoke and the cell population central to the pathogenesis of chronic obstructive pulmonary disease (COPD) and lung cancer. The focus of this study is to identify the differences that two popular alternative nicotine delivery strategies, shisha and electronic cigarettes, have on the airway epithelium compared to cigarette smoking. We hypothesize that both alternative nicotine delivery strategies disorder airway epithelial biology, but in different ways than does cigarette smoking.

DETAILED DESCRIPTION:
Hypothesis and Research Questions We hypothesize that shisha smoking and electronic cigarettes both disorder airway biology, but this disordered biology differs from that resulting from cigarette smoking, suggesting that these alternative nicotine delivery methods will cause lung disease, but perhaps with phenotypes different from that of cigarette smoking.

Aim 1: To assess the hypothesis that shisha smoking disorders the biology of the airway epithelium, but that these changes are distinct from that of cigarette smokers.

Aim 2: To evaluate the hypothesis that when the smoker switches from smoking cigarettes to smoking electronic cigarettes, there is a partial normalization of the disordered airway epithelial biology, but that this partial normalization is different from that associated from complete cessation of cigarette smoking.

Standard and Experimental Procedures

All of the study populations and assessments to be carried out in this protocol are already covered under the IRB approved protocol, "Collection of Airway, Blood and/or Urine Specimens from Subjects for Research Studies" (IRB #1204012331); the only purpose of this protocol is to formalize the timing of assessments so that the underlying hypothesis can be assessed.

The above protocol is designed to assess gene expression in lung cells of nonsmokers, smokers and ex-smokers. The purpose of the present study is to asses if shisha smoking and electronic cigarettes both disorder airway biology, and see if this disordered biology differs from that resulting from cigarette smoking, suggesting that these alternative nicotine delivery methods will cause lung disease, but perhaps with phenotypes different from that of cigarette smoking.

This new protocol will use our existing IRB approved protocol, "Collection of Airway, Blood and/or Urine Specimens from Subjects for Research Studies ("Airway")" (IRB #1204012331), for all of the assessments and procedures of this study. This protocol is designed to formalize the time points at which we carry out the various test parameters (see Table II for a timeline of the study parameters). Recruitment for this protocol will be from the cohort of individuals who are recruited for the "Airway" study. Research subjects recruited into this protocol, will sign both the "Airway" informed consent form and also the consent form for this protocol.

The standard clinical care of our pulmonary physicians is to encourage all smokers to stop smoking; hence, all research participants who smoke will be encouraged to stop smoking. If they decide to do so, they will receive standard of care smoking cessation aids including counseling and medications.

Subjects enrolled in Group E of the study will receive an alternative nicotine delivery method such as electronic cigarettes.

ELIGIBILITY:
Inclusion Criteria:

Group A - Nonsmokers

* All study subjects should be healthy according to the Weill Cornell IRB protocol #1204012331 and be willing and able to provide informed consent for the follow up study with repeated bronchoscopies.
* Subjects will be male and female ≥18 yr of age.
* Nonsmoker is defined as someone who has smoked <100 cigarettes or <10 shisha pipes per lifetime and whose urine nicotine <2 ng/ml and/or urine cotinine <5 ng/ml, at entry into the study.

Group B - Current cigarette smokers

* All study subjects should be healthy according to the Weill Cornell IRB protocol #1204012331 and willing and able to provide informed consent for the follow up study with repeated bronchoscopies.
* Subjects will be male and female ≥18 years of age.
* Active smoker is defined by self-report and urine nicotine >30 ng/ml and/or urine cotinine >50 ng/ml.

Group C - Current shisha smokers

* All study subjects should be healthy according to the Weill Cornell IRB protocol #1204012331 and willing and able to provide informed consent for the follow up study with repeated bronchoscopies.
* Subjects will be male and female ≥18 yr of age.
* Shisha smoker is defined by self-report of smoking >4 pipes/wk and carboxyhemoglobin >2.5.

Group D - Current smokers who stop smoking

* All study subjects should be healthy according to the Weill Cornell IRB protocol #1204012331 and willing and able to provide informed consent for the follow up study with repeated bronchoscopies.
* Subjects will be male and female ≥18 years of age.
* Current smoker is defined by self-report and urine nicotine >30 ng/ml and/or urine cotinine >50 ng/ml.
* Subjects must be a current smoker willing to stop smoking with no contra indications to taking varenicline.

Group E - Current smokers who switch to electronic cigarettes

* All study subjects should be healthy according to the Weill Cornell IRB protocol #1204012331 and willing and able to provide informed consent for the follow up study with repeated bronchoscopies.
* Subjects will be male and female ≥18 years of age. Current smoker is defined by self-report and urine nicotine >30 ng/mL and/or urine cotinine >50 ng/ml.
* Subjects must be willing to switch from tobacco cigarettes to electronic cigarettes.

Exclusion Criteria:

All exclusion criteria apply from the "Airway" (IRB#1204012331) protocol. Additional exclusion criteria specific to this protocol are as follows:

Groups A-E

- No Weill Cornell (including GMS) students will be included, but students from other institutions may be included. A potential pool of Weill Cornell employees may enter this study provided that they are not under the oversight of the study PI or co-investigators.

Groups D and E - Current smokers who stop smoking

- Subjects who are not, in the opinion of the responsible investigator, eligible to take smoking cessation medication due to major depressive and/or other significant psychiatric disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: New York Metropolitan area residents
Sampling Method: Non-Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Number of participants with gene expression changes in the small airway epithelium (SAE) | Study individuals will be enrolled in the study for three months.
  We will measure the effect that shisha smoking has on the small airway epithelium (SAE) by measuring parameters such as the SAE gene expression, DNA methylation, telomere length and cilia length in "pure shisha smokers" (i.e., non-cigarette smokers.) We will compare these parameters to the same parameters measured in non-smokers and cigarette smokers.

SECONDARY OUTCOMES:
Number of participants with gene expression changes in the airway epithelium | Study individuals will be enrolled in the study for three months.
  We will measure the small airway epithelium (SAE) of cigarette smokers who switch to smoking electronic cigarettes by measuring parameters such as the SAE gene expression, DNA methylation, telomere length and cilia length. We will compare these parameters to the same parameters measured in cigarette smokers who stop smoking completely.

CONTACTS AND LOCATIONS:
Overall Officials: Ronald G Crystal, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (2):
- United States (2):
  - Rockefeller University Hospital, New York, New York
  - Weill Cornell Medical College and Weill Cornell Medical Center, Department of Genetic Medicine, New York, New York

IPD SHARING:
Plan to Share IPD: Undecided